CLINICAL TRIAL: NCT02967367
Title: Reliability of Consumer Sleep Trackers in Patients Suffering From Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK/15-06-67/4522
Record Dates: First submitted 2016-09-05; First posted 2016-11-18 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2019-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Jawbone/Withings sleep trackers, Bodymedia Sensewear (Experimental): 2 types of Consumer sleep trackers, including Jawbone and Withings, and one research actigraph (Bodymedia Sensewear) are added to classical polysomnography in order to assess their accuracy to measure sleep parameters in obstructive sleep apnea patients
  Interventions: Device: Jawbone sleep tracker; Device: Withings sleep tracker; Device: BodyMedia Sense Wear accelerometer

INTERVENTIONS:
Device: Jawbone sleep tracker — During one night of polysomnographic recording, investigators are going to place these 3 accelerometers on the wrist of the patient
  Other Names: accelerometer
Device: Withings sleep tracker — During one night of polysomnographic recording, investigators are going to place these 3 accelerometers on the wrist of the patient
Device: BodyMedia Sense Wear accelerometer — During one night of polysomnographic recording, investigators are going to place these 3 accelerometers on the wrist of the patient

SUMMARY:
During last years, numerous sleep trackers have been commercialized. They are intended to give indications about sleep quality/duration in order to give people an internet-based feedback about their own sleep.

For clinical and research purposes, tri-axial accelerometers/multi-sensors devices are used routinely to assess objective sleep quality/patterns. Their use is also validated to estimate sleep in obstructive sleep apnea syndrome (OSA).

The purpose of the present study is to compare the accuracy of consumer-level sleep trackers and validated tools to measure sleep in OSA patients.

DETAILED DESCRIPTION:
During last years, numerous sleep trackers have been commercialized. They are working on accelerometer-based technology. They are intended to give indications about sleep quality/duration in order to give people an internet-based feedback about their own sleep..

For clinical and research purposes, tri-axial accelerometers/multi-sensors devices are used routinely to assess objective sleep quality/patterns. Their use is also validated to estimate sleep in obstructive sleep apnea syndrome (OSA).

The purpose of our study is to compare the accuracy of consumer-level sleep trackers and validated tools to measure sleep in OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* high clinical suspicion of obstructive sleep apnea syndrome

Exclusion Criteria:

* other associated sleep disorder
* inability to sign informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD PhD, Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (1):
- CHu Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
Started | 36
Completed | 22
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time in Bed
Description: time spent in bed during the night (minutes)
Time Frame: one night (up to 600 minutes)
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
Number analyzed (Participants) | 22
min
  PSG | 519 (34)
  Bodymedia Sensewear | 446 (86)
  Jawbone sleep tracker | 522 (45)
  Withings sleep tracker | 524 (122)

2. Primary Outcome: Sleep Efficiency
Description: a percentage corresponding to total sleep time divided by time in bed
Time Frame: one night (up to 600 minutes)
Measure: Mean (Standard Deviation); unit: percentage of time in bed
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
Number analyzed (Participants) | 22
percentage of time in bed
  PSG | 67 (18)
  Bodymedia Sensewear | 80 (14)
  Jawbone sleep tracker | 78 (13)
  Withings sleep tracker | 84 (11)

3. Primary Outcome: Total Sleep Time
Description: time spent sleeping during the night (minutes)
Time Frame: one night (up to 600 minutes)
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
Number analyzed (Participants) | 22
min
  PSG | 344 (92)
  Bodymedia Sensewear | 358 (90)
  Jawbone sleep tracker | 407 (60)
  Withings sleep tracker | 431 (68)

4. Secondary Outcome: Deep Sleep
Description: a percentage corresponding to sleep time spent in deep sleep (stage N3 on polysomnography) divided by total sleep time
Time Frame: one night (up to 600 minutes)
Measure: Mean (Standard Deviation); unit: a percentage of total sleep time
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
Number analyzed (Participants) | 22
a percentage of total sleep time
  PSG | 83 (51)
  Jawbone sleep tracker | 243 (74)
  Withings sleep tracker | 192 (84)

5. Secondary Outcome: Light Sleep
Description: a percentage corresponding to sleep time spent in light sleep (stage N1 and N2 on polysomnography) divided by total sleep time
Time Frame: one night (up to 600 minutes)
Measure: Mean (Standard Deviation); unit: a percentage of total sleep time
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
Number analyzed (Participants) | 22
a percentage of total sleep time
  PSG | 190 (85)
  Jawbone sleep tracker | 163 (69)
  Withings sleep tracker | 239 (54)

ADVERSE EVENTS:
Time Frame: one night, up to 600 minutes
Description: 22 participants were at risk for any adverse events, as usually described
Arm/Group | Jawbone/Withings Sleep Trackers, Bodymedia Sensewear
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT02967367/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT02967367/SAP_001.pdf